CLINICAL TRIAL: NCT00937703
Title: Multicentric Evaluation of Two Telematics Systems (PDA Phone and IVS)in Type 2 Diabetics Patients in Failure of Oral Treatment and Having to Start a Treatment by Basal Insulin, Compared to a Conventional Care. National, Multicentric, Comparative Randomized Study
Brief Title: Multicentric Evaluation of Two Telematics Systems in Type 2 Diabetic Patients in Failure of Oral Treatment and Having to Start Treatment by Basal Insulin
Acronym: TELEDIAB-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008-A00270-55
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2010-03

CONDITIONS: TYPE 2 DIABETES
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group1: Control group (Placebo Comparator): face to face visit à T4mounths
  Interventions: Device: placebo
- Group2: IVS Group (Active Comparator): face to face visit at T4mounths plus telephone visits each 2 weeks
  Interventions: Device: IVS
- Group3: PDAphone group (Active Comparator): PDA system face to face visit at T4mounths plus telephone visits each 2 weeks
  Interventions: Device: PDAphone

INTERVENTIONS:
Device: placebo — paper support for glycaemia face to face visit at T4mounths
  Arms: Group1: Control group
Device: IVS — patients transmit their glycaemia to the IVS, which advises them the insulin amount recommended by their physician in this situation.
  Face to face visit at T4mounths plus telephone visits each 2 weeks.
  Arms: Group2: IVS Group
Device: PDAphone — Patients will receive PDA phone system. They will hace face to face visit at T4mounths and telephone visits each 2 weeks
  Arms: Group3: PDAphone group

SUMMARY:
TELEDIAB-2 is a national, multicenter, controlled, randomised trial. The primary objective of the study is to show that during the initiation of a basal insulin treatment , a computerized decision-making system of adaptation of the insulin, coupled to a distance follow-up (thanks to PDAphone or an interactive vocal server (IVS)), is able to improve metabolic control at the end of 4 mouths as compared with conventional care.

Main judgment criteria: comparison of HbA1c means of the 2 groups profiting from a telemonitoring system compared to the reference group at 4 months.

DETAILED DESCRIPTION:
Secondary objectives :

1. - To compare the 2 methods of telemonitoring employed.
2. - To evaluate the speed of the glycemic attack of the objective to the rising, according to the method of follow-up employed.
3. - To evaluate the satisfaction of the patients and the doctors with respect to systems of telemonitoring, and improvement of the quality of life (DQOL).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes since more than 3 years and claiming a strict balance glycemic;
* Patients treated since at least 3 months, by metformin and secreting insulinic (KNOWN or glinide);
* Patients uncontrolled with HbA1c ≥ 7.5% and < 10% at the inclusion.
* BMI < 40 ;
* Patients requiring a insulin treatment
* Patients agree to start a slow insulin treatment
* Patients already practising the glycemic self-monitoring or agree to learn it and practise it;
* Patients able to include/understand operation and to use the PDA-phone and/or the SVI;
* Patient not taking part in another biomedical research study
* Patients agree to carry out at least 2 finger sticks per day;
* More than 18 years, there is no higher age limit.

Exclusion Criteria:

* Patients introducing any evolutionary pathology associated and not stabilized, exhibitor with an uncontrolled diabetes during the year to come;
* Patients in a situation which justifies of a clinical follow-up diabetologic more frequent than that (quarterly) envisaged by the study
* Patients requiring a transitory passage to insulin;
* Patients needing a hospitalization for the adaptation of insulin doses;
* Patients presenting a cardiologic event
* Patients presenting a hemoglobinopathy interfering with the proportioning of HbA1c;
* Patients suffering from drug-addiction, alcoholism or psychological troubles
* Type 1 or secondary diabetes
* Patients who don't need strict metabolic objectives;
* Pregnant or parturient patients
* person with no freedom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Comparison HbA1c means of the 2 groups profiting from a telemonitoring system compared to the reference group. | To T4 months

SECONDARY OUTCOMES:
Comparison of absolute HbA1c difference | T0-T4 months
Comparison of evolution of HbA1c | T0 and T4 months
Comparison of percentage of patients reaching HbA1c < 7.0% in 4 months | T0 and T4 months
Comparison of percentage of patients within the objective glycemic (the last 3 days Jeun Glycemia average with between 0.73 and 1.08 g/l) at the end of the study, and the average time allowing to achieve this goal | T0 and T4 months
Comparison of the average jeun glycemia the 14 days previous the visit in 4 months | T4 months
Comparison of the frequency of benign hypoglycemias, symptomatic or not, night and severe throughout study | study period
Comparison of the evolution of the weight | T0 and T4 months
Comparison of evolution of the quality of life at the beginning and at the end of the study (the scale of quality of life DHP as well as the items of dimension Satisfaction of the DQOL) | T0 and T4 months
Comparison of the time spent by physicians with patients during visit (either face to face visits or phone call visit); | study period
Comparison of the satisfaction of the patients and physicians with the system and willingness to carry on the use of the system in routine care | 4 months
Effective number of patients carrying on the use of the system in routine care, at their own expense and in agreement with their physician | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CHARPENTIER, MD, Study Chair — Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète; Pierre Yves BENHAMOU, MD PHD, Study Chair — University Hospital, Grenoble
Locations (28):
- France (28):
  - CH Aix en Provence, Aix-en-Provence
  - Centre Hospitalier Intercommunal Alençon-Mamers, Alençon
  - CH Avignon, Avignon
  - Centre Hospitalier de Belfort Montbéliard, Belfort
  - CHU Jean Minjoz, Besançon
  - CHU de Caen, Caen
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CH sud francilien, Corbeil-Essonnes
  - CH de Dreux, Dreux
  - CHU Pierre Zobda-Quitman, Fort de France
  - University Hospital Grenoble, Grenoble
  - CH La Rochelle, La Rochelle
  - CHU de Bicêtre, Le Kremlin-Bicêtre
  - CHU Marseille-Hôpital Nord, Marseille
  - CHU Marseille Hôpitaux Sud, Marseille
  - CH de l'Agglomération Montargoise, Montagis
  - CHU Hôpital Jeanne d'Arc, Nancy
  - CH Nanterre, Nanterre
  - CHU Nantes, Nantes
  - CHU de Nimes, Nîmes
  - Hopital COCHIN, Paris
  - Hopital Haut Leveque, Pessac
  - CHU de Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU de Saint Etienne, Saint-Etienne
  - Hôpital Bégin, Saint-Mandé
  - Centre Hospitalier Strasbourg, Strasbourg
  - Ch Valenciennes, Valenciennes